CLINICAL TRIAL: NCT05177614
Title: A Study to Evaluate the Acceptability of a Multiple Micronutrient-fortified Bouillon Cube in Women and Their Households in Two Districts in the Northern Region of Ghana
Brief Title: Acceptability of Fortified Bouillon Cubes in Northern Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Ghana (Other); Helen Keller International (Other)
Responsible Party: Principal Investigator, Reina Engle-Stone, Ph.D, Assistant Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1687671; 017/12/20 (Other: GHS-ERC)
Record Dates: First submitted 2021-11-06; First posted 2022-01-04 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Food, Fortified; Dietary Habits; Child Development
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: All participants will participate in sensory testing (acceptability, preference and discrimination testing) of three uncooked fortified bouillon cubes (upper-level, lower-level and control), as well as cooked foods containing the three different bouillon cubes. Participants will then be randomized to one of three groups (upper-level, lower-level or control), and receive a 14 day supply of study-provided bouillon cubes to use at home.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper-level multiple micronutrient-fortified bouillon cube (Experimental): 10 gram shrimp-flavoured bouillon cube, consumed ad-lib, fortified with six micronutrients
  Interventions: Dietary Supplement: Upper-level multiple micronutrient-fortified bouillon cube
- Lower-level multiple micronutrient-fortified bouillon cube (Experimental): 10 gram shrimp-flavoured bouillon cube, consumed ad-lib, fortified with six micronutrients
  Interventions: Dietary Supplement: Lower-level multiple micronutrient-fortified bouillon cube
- Control (iodine-fortified bouillon cube) (Placebo Comparator): 10 gram shrimp-flavoured bouillon cube, consumed ad-lib, fortified with one micronutrient
  Interventions: Dietary Supplement: Iodine-fortified bouillon cube

INTERVENTIONS:
Dietary Supplement: Upper-level multiple micronutrient-fortified bouillon cube — 80 µg/g Folic acid 1.2 µg/g Vitamin B12 3 mg/g Zinc (ZnO) 4 mg/g Iron (FePP/citric acid/trisodium citrate) 200 µg/g Vitamin A (retinyl palmitate) 30 µg/g Iodine (KIO3)
  Arms: Upper-level multiple micronutrient-fortified bouillon cube
Dietary Supplement: Lower-level multiple micronutrient-fortified bouillon cube — 28.8 µg/g Folic acid 0.288 µg/g Vitamin B12 1.68 mg/g Zinc (ZnO) 1.3 mg/g Iron (FePP/citric acid/trisodium citrate) 96 µg/g Vitamin A (retinyl palmitate) 30 µg/g Iodine (KIO3)
  Arms: Lower-level multiple micronutrient-fortified bouillon cube
Dietary Supplement: Iodine-fortified bouillon cube — 30 µg/g Iodine (KIO3)
  Arms: Control (iodine-fortified bouillon cube)

SUMMARY:
This study aims to evaluate the acceptability of bouillon cubes fortified with six micronutrients for which deficiency is common among women and children in Ghana and to assess the feasibility and reliability of data collection methods to be used in a planned, more detailed study to evaluate the effect of multiple micronutrient (MN)-fortified bouillon cube on biomarkers of nutrient status, health and development of women and children.

DETAILED DESCRIPTION:
Background: Micronutrient (MN) deficiencies are severe and widespread in West Africa, particularly among young children and women of reproductive age. Bouillon is a promising food fortification vehicle because the product is centrally processed on large scale, consumed by many households in West African countries (even rural, poor households), and consumed by most members of the household in relatively constant amounts. However, several important research questions remain regarding whether the use of fortified bouillon would be feasible, acceptable and effective for preventing micronutrient deficiencies in communities where such deficiencies are common.

Objectives: This study aims (1) to evaluate the acceptability of bouillon cubes formulated with 6 micronutrients for which deficiency is common among women and children in Ghana and (2) to access the feasibility and reliability of data collection methods to be used in a later study of the effects of fortified bouillon, compared to control, on micronutrient status, health, and development.

Methods: This acceptability study will be conducted in the Kumbungu and Tolon districts in the Northern Region, where a recent survey showed that micronutrient deficiencies were common. The investigators will recruit non-pregnant adult women (15+ years old) (n = 84) who are responsible for household meal preparation, to participate in sensory testing of an uncooked fortified bouillon as well as a cooked food containing the fortified bouillon. Subsequently, participants will receive a 14-day supply of fortified bouillon cubes to use at home, after which they will be asked their opinions about the bouillon. Three fortified bouillon formulations will be tested: 1) upper-level bouillon, fortified with iron, zinc, iodine, vitamin A, folic acid, and vitamin B-12, 2) lower-level bouillon, containing the same 6 micronutrients but with lower concentrations of some micronutrients, and 3) a control bouillon, fortified with iodine only. Participants will be in the study for approximately 18 days (study day 0 to study day 17). In addition, children 2-6 years of age in households of enrolled women will be eligible to participate in a pilot study to evaluate the feasibility and test-retest reliability of several methods to assess child development. For these children, child development will be assessed at two home visits during the 14-day period of fortified bouillon use at home.

ELIGIBILITY:
Inclusion Criteria:

Acceptability study:

* self-reported non-pregnant adult women (15+ years)
* responsible for meal preparation in the household
* signed the informed consent form

Child development assessment pilot sub-study:

* 2-6 years of age (24-71 months)
* residing in the same household as an enrolled woman
* child's primary caregiver signs the informed consent form

Exclusion Criteria:

* severe illness warranting immediate hospital referral
* COVID-19 exposure, positive test, or current symptoms (including fever, cough, shortness of breath, loss of smell, vomiting, or diarrhea [> 3 liquid or semi-liquid stools in 24h]) of illness
* chronic severe medical condition (e.g. malignancy) or congenital anomalies requiring frequent medical attention or potentially interfering with nutritional status or affecting child development (children only)
* presence of ailments (such as toothache, or mouth pain) that may impact a participant's ability to complete study activities (women only)
* unable to provide informed consent due to impaired decision making abilities
* current participation in a clinical trial
* reported shrimp, wheat, milk, soy, eggs, celery, fish, or mollusc allergy, or a previous adverse reaction to bouillon by anyone in the household
* refusal to use provided bouillon cubes to prepare household meals while enrolled in the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Sensory perceptions of multiple micronutrient-fortified bouillon cubes (uncooked) | Study day 1
  * centre-based
  * ratings of sensory attributes (appearance, feel, smell, taste and overall) on 5 point hedonic scales
  * ratings of presence of specific organoleptic characteristics ("just-about-right" and "check-all-that-apply)
Sensory perceptions of a soup dish cooked with multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, soup dish randomly assigned to be consumed on study day 1 or 2
  * ratings of sensory attributes (appearance, smell, taste and overall) on 5 point hedonic scales
  * ratings of presence of specific organoleptic characteristics ("just-about-right" and "check-all-that-apply")
Sensory perceptions of a rice-based dish cooked with multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, rice-based dish randomly assigned to be consumed on study day 1 or 2
  * ratings of sensory attributes (appearance, smell, taste and overall) on 5 point hedonic scales
  * ratings of presence of specific organoleptic characteristics ("just-about-right" and "check-all-that-apply")
Ability to discriminate among different multiple micronutrient-fortified bouillon cubes (uncooked) | Study day 1
  * centre-based
  * triangle test (ability to identify the odd sample correctly)
Preference test of multiple micronutrient-fortified bouillon cubes (uncooked) | Study day 1
  * centre-based
  * preference for the multiple micronutrient-fortified bouillon cubes compared to the iodine-fortified control cube (appearance, feel, smell and taste)
Preference test of a soup dish cooked multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, soup dish randomly assigned to be consumed on study day 1 or 2
  * preference for the multiple micronutrient-fortified bouillon cubes compared to the iodine-fortified control cube (appearance, feel, smell and taste) when prepared in commonly consumed dishes
Preference test of a rice-based dish cooked multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, rice-based dish randomly assigned to be consumed on study day 1 or 2
  * preference for the multiple micronutrient-fortified bouillon cubes compared to the iodine-fortified control cube (appearance, feel, smell and taste) when prepared in commonly consumed dishes
Consumption of a soup dish cooked with multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, soup dish randomly assigned to be consumed on study day 1 or 2
  * acceptability of multiple micronutrient-fortified bouillon cubes based on percent of test portions consumed (of commonly consumed dishes cooked with multiple micronutrient-fortified bouillon cubes)
Consumption of a rice-based dish cooked with multiple micronutrient-fortified bouillon cubes | Study day 1 or 2
  * centre-based, rice-based dish randomly assigned to be consumed on study day 1 or 2
  * acceptability of multiple micronutrient-fortified bouillon cubes based on percent of test portions consumed (of commonly consumed dishes cooked with multiple micronutrient-fortified bouillon cubes)
Sensory perceptions of dishes cooked with multiple micronutrient-fortified bouillon cubes | Study day 17
  * in-home acceptability trial (2 weeks), study-provided bouillon cubes used in all household cooking
  * ratings of sensory attributes (appearance, smell, taste and overall) on 5 point hedonic scales
  * ratings of presence of specific organoleptic characteristics ("just-about-right" and "check-all-that-apply")
Quantity of study-provided bouillon cubes used | Study day 17
  * in-home acceptability trial (2 weeks)
  * number of study-provided bouillon cubes used in household over two week trial period
Study-provided bouillon cube use as a proportion of total bouillon use | Study day 17
  * in-home acceptability trial (2 weeks)
  * number of study-provided bouillon cubes used in household over two week trial period, as a proportion of all household bouillon use (study-provided plus non-study provided)
Change in child development scores on the Malawi Developmental Assessment Tool (MDAT) | From study day 3 to study day 17 (2 weeks)
  * gross motor, fine motor, language, and personal-social scores
  * measured twice during study to assess test-retest reliability
  * intraclass correlation coefficient of MDAT
Change in Responsive care and learning opportunities in the home environment: Home Observation for the Measurement of the Environment (HOME) Inventory score | From study day 3 to study day 17 (2 weeks)
  * measured twice during study to assess test-retest reliability
  * intraclass correlation coefficient of HOME inventory

SECONDARY OUTCOMES:
Household-level consumption of salt | Study day 0
  * patterns of salt use prior to the study (pre-intervention)
  * assessed at the initial study visit
Household-level consumption of bouillon | Study day 0
  * patterns of bouillon use prior to the study (pre-intervention)
  * assessed at the initial study visit
Change in willingness to pay for multiple micronutrient-fortified bouillon cubes | Study day 1 and 17
  * assessed pre- and post-intervention
  * hypothetical willingness-to-pay for multiple micronutrient-fortified bouillon cubes before and after exposure to the study-provided bouillon cubes
Themes from focus group discussions | Study day 2 and 17
  * acceptability of the multiple micronutrient-fortified bouillon cubes, experiences of using the multiple micronutrient-fortified bouillon cubes in daily cooking and willingness to use multiple micronutrient-fortified bouillon cubes in the future
  * pre- and post-intervention
  * conducted using a structured focus group discussion guide
Perceived health effects of using study-provided multiple micronutrient-fortified bouillon cubes | Study day 17
  * post-intervention
  * questionnaire to assess perceived positive and negative health effects
Sensory perceptions of dishes cooked with multiple micronutrient-fortified bouillon cubes | Study day 9
  * mid-point of in-home acceptability trial (1 week), study-provided bouillon cubes used in all household cooking
  * ratings of sensory attributes (appearance, smell, taste and overall) on 5 point hedonic scales
  * ratings of presence of specific organoleptic characteristics ("just-about-right" and "check-all-that-apply")

CONTACTS AND LOCATIONS:
Overall Officials: Reina Engle-Stone, PhD, Principal Investigator — University of California, Davis; Seth Adu-Afarwuah, PhD, Principal Investigator — University of Ghana
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
The investigators will commit to Global Access. The investigators intend to 1) publish journal articles describing the study results with an Open Access license, 2) make available information about study methods, such as protocols or standard operating procedures, on the study website, and 3) make available de-identified datasets upon request by the study sponsor or other investigators. Material/DataTransfer Agreements will be developed between study collaborators, sponsor, and any organizations that may request the data; terms of the agreement will be subject to the data handling and storage procedures approved by the University of California, Davis Institutional Review Board (IRB) and Ghana Health Services Ethical Review Committee (GHS-ERC). Organizations that may request the data; terms of the agreement will be subject to the data handling and storage procedures approved by the University of California, Davis IRB and GHS-ERC
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Wessells KR, Kumordzie SM, Becher E, Davis JN, Nyaaba KW, Zyba SJ, Arnold CD, Tan X, Vosti SA, Adams KP, Haskell M, Adu-Afarwuah S, Engle-Stone R. Acceptability of Multiple Micronutrient-Fortified Bouillon Cubes among Women and Their Households in 2 Districts in The Northern Region of Ghana. Curr Dev Nutr. 2023 Dec 8;8(1):102056. doi: 10.1016/j.cdnut.2023.102056. eCollection 2024 Jan. PMID 38304733